CLINICAL TRIAL: NCT01263262
Title: A Comparative Assessment Between Two Surgical Sites of the Rate of Corneal Toxicity and Ototoxicity With the Use of Povidone-iodine Versus Chlorhexidine-alcohol for Facial Lesions Treated With Mohs Micrographic Surgery
Brief Title: A Comparison of Infection Rates Between Two Surgical Sites
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Principal Investigator, Jerry Brewer, Associate Professor of Dermatology, Mayo Clinic
Other Study IDs: 10-004643
Record Dates: First submitted 2010-12-16; First posted 2010-12-20 (Estimated); Last update posted 2013-10-24 (Estimated); Status verified 2013-09

CONDITIONS: Corneal Toxicity; Ototoxicity; Surgical Site Infection
Keywords: Surgical site infection; Corneal toxicity; Ototoxicity; Povidone-iodine; Chlorhexidine-alcohol
MeSH Terms: conditions — Ototoxicity; Surgical Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Does the use of chlorhexidine scrub prior to cutaneous surgery on the face increase the chances of toxicity to the eyes or ears? In addition, does the us eof chlorhexidine scrub on the face prior to cutaneous surgery decrease the chances of a post-operative wound infection?

DETAILED DESCRIPTION:
The intent of this proposed prospective observational cohort study is to determine if there is a difference in the incidence of corneal toxicity and/or ototoxicity in study subjects undergoing Mohs micrographic surgery (MMS) on the face if a povidone-iodine preparation is used pre-operatively as compared to a chlorhexidine-alcohol preparation. It has recently been found that the use of a chlorhexidine-alcohol preparation is superior to the use of a povidone-iodine preparation in preventing post-operative surgical-site infections (SSI) in patients undergoing clean-contaminated surgery. However, the use of chlorhexidine on the face has previously been associated with corneal toxicity and ototoxicity. This study will help to further define previously reported risks of corneal toxicity and ototoxicity associated with the use of a chlorhexidine solution on the face.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing an outpatient cutaneous surgical procedure on the face.

Exclusion Criteria:

* Those who do not consent to participation
* Those undergoing cutaneous surgery for a lesion on the eyelid margin
* Patients with a history of ongoing eye pain
* History of a pre-existing corneal ulcer within 12 months prior to surgery
* History of a perforated tympanic membrane
* Patients with an active infection at the surgical site at the time of surgery.
* If post-operative follow-up is not completed, the study subject will be excluded from the analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive patients 18 years of age or older undergoing Mohs micrographic surgery for a skin neoplasm(s) on the face at the Dermatology Surgery Center at the Mayo Clinic in Rochester, Minnesota, and at the University of Toronto in Toronto, Ontario, Canada, will be included. Exclusion criteria will include: those undergoing MMS for a lesion on the eyelid margin, patients with a history of ongoing eye pain, history of a pre-existing corneal ulcer within 12 months prior to surgery, history of a perforated tympanic membrane, and patients with an active infection at the operative site at the time of surgery. If post-operative follow-up is not completed, the study subject will be excluded from the study.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2011-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Ocular and Ear Toxicities | 1 year
  Comparing ocular and ear toxicities between two institutions with differences in aseptic technique.

SECONDARY OUTCOMES:
Infection rates | 1 year
  compare the infections rates between two institutions with different skin prep practices

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Brewer, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States